CLINICAL TRIAL: NCT02946398
Title: Risk Stratification in Elderly Patients in the Emergency Department
Brief Title: Risk Stratification in the Emergency Department in Acutely Ill Older Patients
Acronym: RiSEuP
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Jacqueline Buijs, Internist, Zuyderland Medisch Centrum
Other Study IDs: NL55867.096.15
Record Dates: First submitted 2016-09-20; First posted 2016-10-27 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Elderly Patiënts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous serum samples: 2. These samples will only be taken in patients who are enrolled in the study in Zuyderland MC (450 patients - anticipated).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elderly patients who visit the ED: elderly patients (65 years and older) who present to the emergency department for internal medicine or gastroenterology

SUMMARY:
Procedures for identification of high-risk elderly patients in the emergency department are lacking.

We aim to identify early risk factors associated with an adverse outcome in elderly patients who visit the emergency department (ED). Second, we aim to find practical tools to identify those elderly patients who are at risk for an adverse outcome in an early stage (by applying and testing triage and risk stratification scores, clinical impression and laboratory results).

With the results of this study, we intend to develop a clinical prediction model to identify older emergency department patients with an increased risk of adverse outcomes.

DETAILED DESCRIPTION:
Background:

Elderly patients (≥65 years of age) constitute an increasing population in emergency departments (EDs) in many countries. These patients are largely different from younger patients and undoubtedly need different approaches in acute care. Commonly used triage systems are not validated in elderly patients. We hypothesize that this factor contributes to a lack of recognition of patients at risk for adverse events or death.

Aim of the study:

* At first, we will try to identify early risk factors associated with adverse outcome such as age, the premorbid state (comorbidity, living status and cognitive/functional state), medication use, vital signs, and number of previous visits to the ED.
* Secondly, we will investigate the discriminating power of several triage and risk stratification scores. In our study, we will retrieve and validate the following triage and risk stratification scores: The Manchester Triage System (MTS) triage score, the Acute Physiology and Chronic Health Evaluation II (APACHE II) score and the Identification of Seniors At Risk-Hospitalised Patients (ISAR-HP) score for all hospitalized patients. Furthermore, we will calculate four well-known disease specific stratification scores: The Glasgow-Blatchford Bleeding (GBS Score) for patients with an upper gastrointestinal bleeding, the Abbreviated Mortality ED Sepsis (abbMEDS) score and Sepsis-related Organ Failure Assessment (SOFA) score and the Confusion, Urea, Respiration, Blood pressure, Age >65 years (CURB-65) score.
* Thirdly, we will investigate the predictive value of the clinical impression of professionals (doctor/nurse) and the disease perception of patient/companion.
* Fourth, we will investigate the predictive value of laboratory tests (routine tests and biomarkers like lactate, N-terminal pro-B-type natriuretic peptide (NT-pro-BNP), high-sensitivity troponin (hs-TnT), procalcitonin (PCT) and d-dimer.
* At last, we intend to develop a clinical prediction model for short-term mortality and test the predictive ability of this model for the other adverse outcomes/endpoints. This model will be validated in an external cohort.

Study procedure:

The design is a multi-center prospective observational cohort study. The study will take place in Zuyderland MC in Heerlen and Maastricht UMC+ in the Netherlands. On presentation to the ED the patients will be given information about the study and informed consent will be signed. The patient or family member/companion, the nurse and the doctor will be asked to fill out a questionnaire in the ED (5 questions for patient/family and 9 questions for doctor or nurse). These questions will be used for evaluation of the clinical impression of the doctor/nurse and disease perception by the patient/companion. At the ED, 2 extra venous samples and one arterial blood gas sample will be taken in patients participating in the study in Zuyderland M.C. Blood gas analysis will take place immediately and the results will be presented to the attending doctor. Analysis of the biomarkers from the venous blood samples will take place after a few weeks and the results will be blinded in this study. Routine laboratory test will be analyzed in both hospitals. During the days and weeks after inclusion, data will be obtained from patients medical records. During the days and weeks after inclusion, data will be obtained from patients medical records. All patients will be followed up for 30 days and if possible for one year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Visit to the emergency department for the internist/gastroenterologist
* Informed consent

Exclusion Criteria:

* Earlier participation in study (patients can only be included once)
* No informed consent
* Inability to speak Dutch or English
* Admission to a ward of another specialty than internal medicine/gastroenterology

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients ≥65 years of age who present to the ED for internal medicine or gastroenterology within the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2019-07-06 (Actual)

PRIMARY OUTCOMES:
30-day all cause mortality | 30 days
  all cause mortality within 30 days (both in- and out-hopsital)

SECONDARY OUTCOMES:
composite secondary outcome | 30 days or 30 days after hospital discharge
  1. Length of hospital stay longer than 1 week
  2. ICU/MCU admission
  3. all cause mortality within 30 days of presentation to the ED
  4. Readmission within 30 days of discharge from the hospital
  5. Discharge to another residence than previous address (nursing home/hospice)
all cause mortality after 1 year | 1 year
  all cause mortality after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Buijs, dr., Principal Investigator — Zuyderland M.C.
Locations (2):
- Netherlands (2):
  - Zuyderland Medisch Centrum, Heerlen, Limburg
  - Maastricht UMC+, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zelis N, Hundscheid R, Buijs J, De Leeuw PW, Raijmakers MT, van Kuijk SM, Stassen PM. Value of biomarkers in predicting mortality in older medical emergency department patients: a Dutch prospective study. BMJ Open. 2021 Jan 31;11(1):e042989. doi: 10.1136/bmjopen-2020-042989. PMID 33518523
- [Derived] Zelis N, Huisman SE, Mauritz AN, Buijs J, de Leeuw PW, Stassen PM. Concerns of older patients and their caregivers in the emergency department. PLoS One. 2020 Jul 9;15(7):e0235708. doi: 10.1371/journal.pone.0235708. eCollection 2020. PMID 32645113
- [Derived] Zelis N, Buijs J, de Leeuw PW, van Kuijk SMJ, Stassen PM. Study protocol for a multicentre prospective cohort study to identify predictors of adverse outcome in older medical emergency department patients (the Risk Stratification in the Emergency Department in Acutely Ill Older Patients (RISE UP) study). BMC Geriatr. 2019 Mar 4;19(1):65. doi: 10.1186/s12877-019-1078-2. PMID 30832571